CLINICAL TRIAL: NCT00004444
Title: Pilot Randomized Study of Paromomycin (Aminosidine) vs Streptomycin for Uncomplicated Pulmonary Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: University of Illinois at Chicago (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13445; UIC-FDR001167
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: bacterial infection; immunologic disorders and infectious disorders; mycobacterium infection; mycobacterium tuberculosis infection; rare disease
MeSH Terms: conditions — Tuberculosis, Pulmonary; Bacterial Infections; Immune System Diseases; Communicable Diseases; Mycobacterium Infections; Tuberculosis; Rare Diseases | interventions — Paromomycin; Streptomycin

INTERVENTIONS:
Drug: paromomycin
Drug: streptomycin

SUMMARY:
OBJECTIVES: I. Compare the pharmacokinetics and early bactericidal activity of paromomycin (aminosidine) vs streptomycin for the treatment of uncomplicated pulmonary tuberculosis.

II. Compare the tolerability of these two drugs in these patients. III. Establish the relationships between achieved serum concentration, minimal inhibitory concentration, and early bactericidal activity of paromomycin and streptomycin.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are randomized to one of three treatment arms. Patients in arms I and II receive one of two doses of paromomycin intramuscularly once a day for 3 days. Patients in arm III receive streptomycin intramuscularly once a day for 3 days. All patients then begin a course of standard therapy for tuberculosis.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Microbiologically proven uncomplicated pulmonary tuberculosis Positive direct sputum smear for acid-fast bacilli OR Presumptive diagnosis based on clinical and radiological findings
* No known risk factors for multidrug resistant tuberculosis (MDR TB) including: Domicile, shelter, or prison exposure to MDR TB within 6 months Residence in a specific domicile, shelter, or prison cell block within 6 months of a known outbreak of MDR TB Hospitalization, within 6 months, on a medical service or unit in which nosocomial transmission of MDR TB is known to have occurred
* No clinical evidence of CNS or miliary tuberculosis
* HIV seronegative

--Prior/Concurrent Therapy--

* Biologic therapy: At least 12 weeks since immune modulators (including colony-stimulating factors, interferons, or interleukins)
* Chemotherapy: No concurrent chemotherapy
* Endocrine therapy: At least 12 weeks since corticosteroids
* Other: At least 2 years since treatment or prophylaxis for tuberculosis At least 12 weeks since treatment with any drug with activity against tuberculosis, including: All standard drugs used for tuberculosis Clofazimine Rifabutin Quinolones Aminoglycosides At least 12 weeks since pentoxifylline

--Patient Characteristics--

* Hematopoietic: Absolute neutrophil count at least 1,000/mm3
* Renal: Creatinine clearance greater than 60 mL/min
* Pulmonary: No chronic obstructive pulmonary disease
* Other: Not pregnant Fertile patients must use effective contraception No history of intolerance or known hypersensitivity to aminoglycosides No known or suspected Mycobacterium avium complex infection No other serious, acute infection No diabetes No major organ dysfunction No malignancy requiring chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1994-11; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Paul Kanyok, Study Chair — University of Illinois at Chicago